CLINICAL TRIAL: NCT01666951
Title: Ph 2 Double-blind, Double-dummy, Multicenter, Prospective, Rand Study of PK of LCP-Tacro™ Tablets Once Daily, Compared to Prograf® Caps, Twice Daily, for Prevention of Acute Allograft Rejection in De Novo Adult Kidney Transplant Recipients
Brief Title: Multicenter, Prospective, Rand, PK Study of LCP-Tacro™ Compared to Prograf® Capsules in De Novo Adult Kidney Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LCP-Tacro 2019
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Results first posted 2015-07-07 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-06

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCP-Tacro (Experimental): LCP-Tacro Tablets, once daily (Veloxis Pharmaceuticals A/S, Horsholm, DK)
  Interventions: Drug: LCP-Tacro tablets
- Prograf (Active Comparator): Prograf Capsules, twice daily (Astellas Pharma US, Deerfield, IL)
  Interventions: Drug: Prograf

INTERVENTIONS:
Drug: LCP-Tacro tablets — Tacrolimus
  Other Names: Prograf
  Arms: LCP-Tacro
Drug: Prograf — Tacrolimus
  Other Names: Prograf Capsules twice daily
  Arms: Prograf

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of LCP-Tacro tablets administered once-daily compared to Prograf capsules administered twice-daily after kidney transplantation.

DETAILED DESCRIPTION:
This is a 2-arm , parallel group, prospective, double-blind, double-dummy, multicenter,clinical trial to evaluate the pharmacokinetics of LCP-Tacro tablets once daily in comparison to Prograf capsules twice-daily after kidney transplantation.

ELIGIBILITY:
Inclusion criteria

* Give written consent
* Male and female subjects between the ages of 18 and 70 years, inclusive
* Must be receiving primary or secondary renal allograft from a deceased donor or non- HLA identical living donor
* WOCBP must have a negative pregnancy test
* Must have negative cross-match test and be ABO-compatible
* Must be able to swallow tablets and capsules

Exclusion criteria

* Recipients of any previous nonrenal or concurrent transplant
* Have panel reactive antibody >50%
* Any condition that may affect study drug absorption BMI <18 kg/m2 or > 45 kg/m2
* History of alcohol abuse with less than 6 months of sobriety
* History of recreational drug abuse with less than 6 months of documented abstinence
* Screening 12-lead ECG demonstrating CS abnormalities (including QTc prolongation)
* WOCBP and are either pregnant, lactating, planning to become pregnant or with a positive serum or urine pregnancy test
* Subjects (male or female) with reproductive potential who are unwilling/unable to use a double-barrier method
* Oral temperature (prior to study drug dosing) of 38.0ºC or higher
* CS active infections (eg, those requiring hospitalization, or as judged by the Investigator)
* Known hereditary immunodeficiency
* Malignancies or with a history of malignancies (within the last 5 years) with the exception of local, noninvasive, fully excised cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, or cervical carcinoma in situ
* Expect to receive within 2 months after randomization, or have received within 3 months prior to screening, any of the following: sirolimus, everolimus, belatacept, or cyclophosphamide
* Any psychiatric or medical condition that, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
* Clinically symptomatic CHF or documented EJF of less than 45%
* Significant COPD, pulmonary restrictive disease or significant pulmonary hypertension
* Enrolled in another investigational drug or device study, or who are less than 30 days since discontinuing
* Laboratory variables that are abnormal (outside laboratory reference range) and CS
* Positive results of any of the following serological tests: human immunodeficiency virus (HIV)-1 antibody, hepatitis B virus (HBV) surface antigen (HBsAg), anti-hepatitis B core antibody (HBcAb), and anti-hepatitis C virus (HCV) antibody (HCV Ab)
* Subjects who have had primary focal segmental glomerulosclerosis
* Donor parameters must not include any of the following known conditions:

Donor with positive serological test result for HIV-1, HBV or HCV Donor with history of malignant disease (current or historical) Cold ischemia time >30 hours Non-heart-beating donor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Polvino, MD, Study Director — Veloxis Pharmaceuticals
Locations (13):
- United States (13):
  - Clinical Investigative Site 000015, San Diego, California
  - Clinical Investigative Site 000012, San Francisco, California
  - Clinical Investigative Site 00004, Aurora, Colorado
  - Clinical Investigative Site 000002, Tampa, Florida
  - Clinical Investigative Site 000005, Lexington, Kentucky
  - Clinical Investigative Site 000009, Ann Arbor, Michigan
  - Clinical Investigative Site 000010, Livingston, New Jersey
  - Clinical Investigative Site 000011, Buffalo, New York
  - Clinical Investigative Site 00006, New York, New York
  - Clinical Investigative Site 00008, Cleveland, Ohio
  - Clinical Investigative Site 00003, Philadelphia, Pennsylvania
  - Clinical Investigative Site 000013, Dallas, Texas
  - Clinical Investigative Site 00001, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LCP-Tacro | Prograf
Started | 18 | 18
Completed | 17 | 17
Not Completed | 1 | 1
Not completed — Not dosed | 1 | 1

BASELINE CHARACTERISTICS:
Population: The two patients that were randomized but not does (one in eacj treatment arm) are not included in the demographics
Groups:
- Total: Total of all reporting groups
Arm/Group | LCP-Tacro | Prograf | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (13.92) | 46.4 (11.49) | 49.0 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 14 | 9 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 16 | 13 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 10 | 12 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Daytime, Nighttime and Overnight Systolic Blood Pressure (SBP) on Day 14.
Description: At selected sites, a 24-hour measurement of blood pressure will be performed to assess the variability (ei, "nighttime dipping") between the two Groups at Days 14.
Time Frame: 14 days
Population: 18 patients participated in the 24-hour blood pressure assessment, 8 in the LCP-Tacro arm and 10 on the Prograf arm.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCP-Tacro | Prograf
Number analyzed (Participants) | 8 | 10
mmHg
  Daytime SBP | 140.96 (10,311) | 131.54 (13.835)
  Nighttime SBP | 140.69 (9.147) | 133.38 (17.875)
  Overnight SBP | 140.80 (10.347) | 132.54 (18.127)

2. Other Pre Specified Outcome: Daytime, Nighttime Overnight Systolic Blood Pressure (SBP) on Day 28.
Description: At selected sites, a 24-hour measurement of blood pressure will be performed to assess the variability (ei, "nighttime dipping") between the two Groups at Day 28.
Time Frame: 28 days
Population: 18 patients participated in the 24-hour blood pressure assessment, 8 in the LCP-Tacro arm and 10 on the Prograf arm.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCP-Tacro | Prograf
Number analyzed (Participants) | 8 | 10
mmHg
  Daytime SBP | 139.05 (14.722) | 130.84 (15.754)
  Nighttime SBP | 137.18 (13.283) | 129.09 (16.447)
  Overnight SBP | 136.11 (13.539) | 127.70 (16.599)

3. Primary Outcome: Pharmacokinetics (AUC) of LCP-Tacro Compared to Prograf After Kidney Transplantation
Description: The pharmacokinetic parameter (AUC) was evaluated on Day 1 in adult de novo kidney recipients. Samples were collected from 0 to 24 hours post dose.
Time Frame: 1 days
Population: The PK assessments were performed on the PK populations set which consists of 26 patients, 14 of whom received LCP-Tacro and 12 of whom who received Prograf.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | LCP-Tacro | Prograf
Number analyzed (Participants) | 14 | 12
ng*hr/mL | 382.72 (233.84) | 147.82 (85.31)

4. Primary Outcome: Pharmacokinetics (AUC) of LCP-Tacro Compared to Prograf After Kidney Transplantation
Description: The pharmacokinetic parameter (AUC) was evaluated on Day 14 in adult de novo kidney recipients. Samples were collected from 0 to 24 hours post dose.
Time Frame: 14 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | LCP-Tacro | Prograf
Number analyzed (Participants) | 14 | 12
ng*hr/mL | 371.43 (133.85) | 244.63 (66.92)

5. Primary Outcome: Pharmacokinetics (AUC) of LCP-Tacro Compared to Prograf After Kidney Transplantation
Description: The pharmacokinetic parameter (AUC) was evaluated on Day 28 in adult de novo kidney recipients. Samples were collected from 0 to 24 hours post dose.
Time Frame: 28 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | LCP-Tacro | Prograf
Number analyzed (Participants) | 14 | 12
ng*hr/mL | 357.39 (146.64) | 205.79 (36.25)

6. Primary Outcome: Pharmacokinetics (Cmax and C24) of LCP-Tacro Compared to Prograf After Kidney Transplantation
Description: The pharmacokinetic parameter (Cmax and C24) was evaluated on Day 1 in adult de novo kidney recipients.
Time Frame: 1 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LCP-Tacro | Prograf
Number analyzed (Participants) | 14 | 12
ng/mL
  Cmax | 32.68 (20.51) | 12.97 (7.08)
  C24 | 13.32 (8.89) | 5.72 (5.28)

7. Primary Outcome: Pharmacokinetics (Cmax and C24) of LCP-Tacro Compared to Prograf After Kidney Transplantation
Description: The pharmacokinetic parameter (Cmax and C24) was evaluated on Day 14 in adult de novo kidney recipients.
Time Frame: 14 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LCP-Tacro | Prograf
Number analyzed (Participants) | 12 | 14
ng/mL
  Cmax | 30.08 (14.27) | 18.98 (6.59)
  C24 | 9.11 (2.86) | 7.54 (2.50)

8. Primary Outcome: Pharmacokinetics (Cmax and C24) of LCP-Tacro Compared to Prograf After Kidney Transplantation
Description: The pharmacokinetic parameter (Cmax and C24) was evaluated on Day 28 in adult de novo kidney recipients.
Time Frame: 28 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LCP-Tacro | Prograf
Number analyzed (Participants) | 12 | 14
ng/mL
  Cmax | 32.51 (18.74) | 17.38 (4.07)
  C24 | 9.31 (3.44) | 6.75 (2.22)

9. Primary Outcome: Pharmacokinetics (Tmax) of LCP-Tacro Compared to Prograf After Kidney Transplantation
Description: The pharmacokinetic parameter (Tmax) was evaluated on Day 1 in adult de novo kidney recipients.
Time Frame: 1 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | LCP-Tacro | Prograf
Number analyzed (Participants) | 14 | 12
hour | 11.26 (7.49) | 7.39 (6.37)

10. Primary Outcome: Pharmacokinetics (Tmax) of LCP-Tacro Compared to Prograf After Kidney Transplantation
Description: The pharmacokinetic parameter (Tmax) was evaluated on Day 14 in adult de novo kidney recipients.
Time Frame: 14 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | LCP-Tacro | Prograf
Number analyzed (Participants) | 14 | 12
hour | 7.03 (5.69) | 5.03 (5.81)

11. Primary Outcome: Pharmacokinetics (Tmax) of LCP-Tacro Compared to Prograf After Kidney Transplantation
Description: The pharmacokinetic parameter (Tmax) was evaluated on Day 28 in adult de novo kidney recipients.
Time Frame: 28 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | LCP-Tacro | Prograf
Number analyzed (Participants) | 14 | 12
hour | 5.69 (4.11) | 7.69 (6.87)

12. Primary Outcome: Pharmacokinetics (Fluctuation) of LCP-Tacro Compared to Prograf After Kidney Transplantation
Description: The pharmacokinetic parameter (Fluctuation) was evaluated on Day 14 in adult de novo kidney recipients.
Time Frame: 14 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of fluctuation
Arm/Group | LCP-Tacro | Prograf
Number analyzed (Participants) | 14 | 12
Percentage of fluctuation | 126.86 (57.65) | 114.73 (52.36)

13. Primary Outcome: Pharmacokinetics (Fluctuation) of LCP-Tacro Compared to Prograf After Kidney Transplantation
Description: The pharmacokinetic parameter (Fluctuation) was evaluated on Day 28 in adult de novo kidney recipients.
Time Frame: 28 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of fluctuation
Arm/Group | LCP-Tacro | Prograf
Number analyzed (Participants) | 14 | 12
Percentage of fluctuation | 144.78 (84.63) | 131.4 (75.96)

14. Other Pre Specified Outcome: Ratio of Nighttime to Daytime Systolic Blood Pressure (SBP) on Day 14.
Description: as for outcome 1
Time Frame: 14 days
Population: 18 patients participated in the 24-hour blood pressure assessment, 8 in the LCP-Tacro arm and 10 on the Prograf arm.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | LCP-Tacro | Prograf
Number analyzed (Participants) | 8 | 10
ratio
  Night:Day ratio SBP | 0.99 (0.035) | 1.01 (0.057)
  Overnight:Day Ratio SBP | 1.00 (0.053) | 1.01 (0.057)

15. Other Pre Specified Outcome: Ratio of Nighttime to Daytime Systolic Blood Pressure (SBP) on Day 28.
Description: At selected sites, a 24-hour measurement of blood pressure will be performed to assess the variability (ei, "nighttime dipping") between the two Groups at Days 28.
Time Frame: 28 days
Population: 18 patients participated in the 24-hour blood pressure assessment, 8 in the LCP-Tacro arm and 10 on the Prograf arm.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | LCP-Tacro | Prograf
Number analyzed (Participants) | 8 | 10
ratio
  Night:Day ratio SBP | 0.99 (0.035) | 0.98 (0.067)
  Overnight:Day Ratio SBP | 0.99 (0.064) | 0.98 (0.067)

16. Other Pre Specified Outcome: Evaluation of the Short-term Efficacy of LCP-Tacro After the Start of Dosing.
Description: The efficacy is measured by the number of treatment failures defined as all-cause mortality, Graft Failure, Biopsy Proven Acute Rejection (BPAR) and Lost to follow up.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | LCP-Tacro | Prograf
Number analyzed (Participants) | 18 | 16
participants
  All-cause mortality | 0 | 0
  Graft Failure | 0 | 0
  BPAR | 2 | 0
  Lost to follow up | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of study drug and until 30 days after last dose of study drug for at total of 2 months.
Arm/Group | LCP-Tacro | Prograf
Serious Adverse Events (participants affected / at risk) | 5/17 | 5/17
Other Adverse Events (participants affected / at risk) | 17/17 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCP-Tacro (N=17) | Prograf (N=17)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrilation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 2 (2) | 0 (0)
Pelvic Abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Renal INjury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCP-Tacro (N=17) | Prograf (N=17)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrilation (Cardiac disorders) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Catheter site realted reaction (General disorders) | 1 (1) | 0 (0)
Exercise tolerance decreased (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Oral Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Vulvovaginal myotic infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 3 (3) | 3 (3)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Drug level increased (Investigations) | 1 (1) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Polyomavirus test positive (Investigations) | 1 (2) | 0 (0)
Vitamin D decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypovitaminosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Vimatin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 4 (4) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Perinephric effusion (Nervous system disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 4 (4)
Hypotension (Vascular disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other